CLINICAL TRIAL: NCT05227859
Title: Assessment of the Effects of Piezocision and Low-level Laser Therapy on Orthodontic Tooth Movement During Canine Retraction and the Associated Dentoalveolar Changes: A Three-arm Randomized Controlled Clinical Trial
Brief Title: Which is Better Piezosurgery or LLLT in Accelerating Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-01-2022
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Class II Malocclusion
Keywords: LLLT; Piezocision; Canine retraction; Acceleration
MeSH Terms: conditions — Overbite | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Piezocision therapy (Experimental): In this group of patients, the canine will be retracted in association with piezocision.
  Interventions: Procedure: Piezocision
- Low-level laser therapy (Experimental): In this group of patients, the canine will be retracted in association with LLLT.
  Interventions: Device: Low-level laser
- Conventional treatment (Active Comparator): In this group of patients, the canine will be retracted conventionally without any acceleration intervention.
  Interventions: Device: Conventional treatment

INTERVENTIONS:
Procedure: Piezocision — After anesthesia, three vertical incisions will be made (3-mm depth and 8-10 mm length) mesial and distal the upper canine as well as at an equal distance from the upper canine and 2nd premolar. The surgical procedures will be repeated after six weeks (only the mesial and distal canine incisions will be done)
  Arms: Piezocision therapy
Device: Low-level laser — GaALAs diode laser (wavelength: 810 nm and exposure time of 10 seconds\point) will be applied around the upper canine in 10 sites from buccal and palatal. The middle of the extraction site will be also irradiated in 4 sites (2 buccally and 2 palatally). The LLLT will be applied 5 times in the first month of canine retraction, then every two weeks until class I canine relationship will be achieved.
  Arms: Low-level laser therapy
Device: Conventional treatment — The upper canine destalization will be done using NiTi springs. The force level will be controlled every 2 weeks. Retraction will be stopped when a class I canine relationship in both sides.
  Arms: Conventional treatment

SUMMARY:
Sixty patients requiring extraction-based treatment of the maxillary first premolars, followed by retraction of the maxillary canines, will be randomly assigned to three groups: piezocision, low-level laser therapy, and control. In each group, canine retraction will be initiated after completion of the leveling and alignment phase, using closed nickel-titanium coil springs that apply 150 g of force per side. For anchorage, a soldered transpalatal arch will be used.

Pre- and post-distalization dental casts will be assessed to evaluate the rate of canine retraction, canine rotation, and anchorage loss over the follow-up period until a Class I canine relationship is achieved. Periodontal health will be assessed before and after canine retraction by evaluating the following parameters: plaque index, gingival index, bleeding index, and probing depth.

DETAILED DESCRIPTION:
Before enrollment of each subject in the study, they will undergo a comprehensive assessment to ensure their eligibility. The operator will inform them of the study's aim and request written informed consent.

At the end of the leveling and alignment stage, the upper first premolars will be extracted. The rectangular stainless steel archwires (0.019" × 0.025") will be inserted, and after one month, canine retraction will be initiated.

Regarding the Piezocision, after anesthesia, three vertical incisions will be made (3-mm depth and 8-10 mm length) mesial and distal to the upper canine, as well as at an equal distance from the upper canine and the 2nd premolar. The surgical procedures will be repeated after six weeks (only the mesial and distal canine incisions will be done) Regarding low-level laser therapy (LLLT), a GaAlAs diode laser (wavelength: 810 nm; exposure time: 10 seconds per point) will be applied around the upper canine at 10 sites, buccally and palatally. The central portion of the extraction site will also be irradiated at four sites (2 buccally and two palatally). LLLT will be applied 5 times during the first month of canine retraction, then every 2 weeks until a Class I canine relationship is achieved.

The upper canine destalization will be done using NiTi springs. The force level will be controlled every 2 weeks. Retraction will be stopped when a class I canine relationship is present on both sides.

Dental casts will be used to quantify the anteroposterior movement of the upper canines and first molars at 30-day intervals until the Class I canine relationship is achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 17-28 years.
2. Class II Division 1 malocclusion :

   * Mild/moderate skeletal Class II (sagittal discrepancy angle ≤7)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles: mandibular/cranial base angle, maxillary/mandibular plane angle, and facial axis angle)
   * Mild to moderate crowding ≤ 4
3. Permanent occlusion.
4. Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs), …)
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
5. Patient had previous orthodontic treatment

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-08 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Duration of upper canine retraction | The months required to complete the retraction procedure will be recorded. Completion of this procedure is expected to occur within four months in the experimental groups and seven months in the control group
  Assessment will be performed by calculating the months required to achieve complete retraction of the upper canine retraction through clinical examination.
Rate of retraction | Time Frame: The calculation of the rate of retraction will be done once the retraction procedures have finished. Completion of this procedure is expected to occur within 4 months in the experimental groups and 7 months in the control group.
  Assessment will be performed on study models. The amount of distance being retracted in millimeters will be divided by the duration of retraction in weeks to give an estimation of the retraction rate.

SECONDARY OUTCOMES:
Change in Molars' positions | T0: 1 day before the beginning of canine retraction; T1: after 1 month of retraction; T2: after 2 months of retraction; T3: after 3 months; and T4: at the end of retraction (expected to be within 4 months to 7 months))
  The amount of distance being traveled by the first molars is going to be measured on study models taken at monthly intervals until the end of the retraction phase.
Change in canine' rotation | T0: 1 day before the beginning of canine retraction; T1: after 1 month of retraction; T2: after 2 months of retraction; T3: after 3 months of retraction; and T4: at the end of retraction (expected to be within 4 months to 7 months)
  The amount of the rotation of canine is going to be measured on study models taken at monthly intervals until the end of the retraction phase.
Change in the plaque index | T0: immediately before the commencement of the retraction phase; T1: at the end of the retraction phase, which is expected to occur within 4 months in the experimental groups and 7 months in the control group
  Assessment will be performed using a gingival probe to evaluate oral hygiene status in enrolled patients.
  A. (0) = No plaque. B. (1) = A film of plaque stuck to the free gingival margin and adjacent area of the tooth.
  C. (2) = Moderate accretion of soft deposits on the tooth and gingival margin or within the gingival pocket.
  D. (3) = Abundance of soft material on the tooth and gingival margin and/or within the gingival pocket.
Change in the gingival index | T0: immediately before the commencement of the retraction phase; T1: at the end of the retraction phase, which is expected to occur within 4 months in the experimental groups and 7 months in the control group
  Assessment will be achieved using a gingival probe to assess the status of the gingival tissues around the upper teeth (from the 2nd premolar to the contralateral 2nd premolar).
  A. (0) = Normal gingiva. B. (1) = Mild inflammation: minor color change, slight oedema. No bleeding on probing.
  C. (2) = Moderate inflammation: redness, oedema, glazing, and bleeding on probing.
  D. (3) = Severe inflammation: marked redness and oedema, ulceration, and tendency to spontaneous bleeding.
Change in the papillary bleeding index | T0: immediately before the commencement of the retraction phase; T1: at the end of the retraction phase, which is expected to occur within 4 months in the experimental groups and 7 months in the control group
  Assessment will be achieved using a gingival probe to assess the status of periodontal tissues around the upper teeth (from the 2nd premolar to the contralateral 2nd premolar).
  A. (0) = No bleeding. B. (1) = A single, discrete bleeding point appears. C. (2) = Several isolated bleeding points or a single fine line of blood appears.
  D. (3) = The interdental triangle fills with blood shortly after probing. E. (4) = Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.
Change in the probing depth | T0: immediately before the commencement of the retraction phase; T1: at the end of the retraction phase, which is expected to occur within 4 months in the experimental groups and 7 months in the control group
  Assessment will be achieved using a gingival probe. It will be measured clinically as the distance from the free gingival margin to the gingival sulcus around the six maxillary anterior teeth and 2nd premolars.

CONTACTS AND LOCATIONS:
Overall Officials: Doa'a Tahseen Alfailany, DDS, Principal Investigator — Department of Orthodontics, University of Damascus Dental School, Syria; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Professor of Orthodontics, University of Damascus Dental School, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdelhameed AN, Refai WMM. Evaluation of the Effect of Combined Low Energy Laser Application and Micro-Osteoperforations versus the Effect of Application of Each Technique Separately On the Rate of Orthodontic Tooth Movement. Open Access Maced J Med Sci. 2018 Nov 15;6(11):2180-2185. doi: 10.3889/oamjms.2018.386. eCollection 2018 Nov 25. PMID 30559886
- [Background] Rajasekaran UB, Krishna Nayak US. Effect of prostaglandin E1 versus corticotomy on orthodontic tooth movement: an in vivo study. Indian J Dent Res. 2014 Nov-Dec;25(6):717-21. doi: 10.4103/0970-9290.152170. PMID 25728102
- [Background] Turker G, Yavuz I, Gonen ZB. Which method is more effective for accelerating canine distalization short term, low-level laser therapy or piezocision? A split-mouth study. J Orofac Orthop. 2021 Jul;82(4):236-245. doi: 10.1007/s00056-020-00250-6. Epub 2020 Sep 29. PMID 32990775
- [Background] Cagli Karci I, Baka ZM. Assessment of the effects of local platelet-rich fibrin injection and piezocision on orthodontic tooth movement during canine distalization. Am J Orthod Dentofacial Orthop. 2021 Jul;160(1):29-40. doi: 10.1016/j.ajodo.2020.03.029. Epub 2021 May 4. PMID 33962809
- [Background] Abbas NH, Sabet NE, Hassan IT. Evaluation of corticotomy-facilitated orthodontics and piezocision in rapid canine retraction. Am J Orthod Dentofacial Orthop. 2016 Apr;149(4):473-80. doi: 10.1016/j.ajodo.2015.09.029. PMID 27021451